CLINICAL TRIAL: NCT05305937
Title: Implantation of CEST and CESL MRI Methods for Detection of Breast Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Rotem Sivan-Hoffmann, Head of Radiology department, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0201-21
Record Dates: First submitted 2022-02-23; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Malignant Tumor of Breast; Benign Breast Lumps; High-Risk Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- One arm - all patients (Experimental)
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — All patients will be scanned twice during the same MRI session, before and 2 hours after taking glucosamine orally. In addition to the CEST scans with glucosamine, patients will undergo MRI scans with the standard contrast agent of gadolinium. This procedure will be done following the CEST scan

SUMMARY:
MRI is a well-established method in breast imaging. It gives excellent morphological information but does not reflect the metabolic activity leading to high proportion of false positive results. PET-CT fulfills this gap but suffers from low resolution and the risk of radiation damage. Lately, chemical exchange saturation transfer (CEST) MRI of glucose has been proposed as a new molecular imaging approach for diagnosing tumors given its high sensitivity at the molecular level and the known enhanced glucose uptake by tumors. Several glucose analogs were examined as possible candidates for imaging of breast tumors. One of the most promising agent for CEST-MRI is glucosamine (GlcN); owing to its phosphorylated products that accumulate in breast tumors, it enables to reflect their metabolic profile. In preclinical experiments glucosamine exhibits enhanced CEST signals in 4T1 and MCF7 implanted breast cancer cells in mice. Its potential for the human clinical application is strengthened by its lack of toxicity. Here the investigators propose to test the method for human subjects on a clinical MRI setup. The goal of this study is to develop innovative molecular imaging modality based on CEST-MRI of GlcN for the detection of breast tumors. The investigators will use the newly developed CEST-MRI modality for the detection of benign and malignant breast cancer in a clinical MRI scanner.

.

DETAILED DESCRIPTION:
The primary aim of this study is to develop innovative molecular imaging modality based on the chemical exchange saturation transfer MRI (CEST-MRI) of glucosamine (GlcN) to visualize and measure breast tumors. GlcN has been shown to have good breast tumor targeting properties allowing its detection in laboratory animals under CEST MRI technique. The investigators will use the newly developed CEST-MRI modality for the detection of benign and malignant breast cancer in a clinical MRI scanner

STUDY AIMS

1. Investigate the possibility of obtaining a new contrast image of breast cancer tumors using glucosamine as a new contrast agent using the CEST imaging method (Chemical Exchange Saturation Transfer chemical exchange during saturation transition) and/or the CESL (Spin Lock chemical exchange method).
2. A comparison of the contrast image obtained by the novel GlcN CEST-MRI and/or CESL-MRI methods to that obtained by traditional MRI methods like T1, T2.
3. Using the GlcN- CEST-MRI / or CESL-MRI approaches, compare the signal obtained by malignant and benign tumors, examination if these methods can distinguish between the two types of tumors.

Patients bearing solid breast tumors will be scanned at the clinical MRI setup. The scans will include short anatomical scans (of T1 and T2 images) and CEST imaging. Patients will be required to fast for at least 4 hours before the scan (can drink water during fasting). The participants will be asked to drink glucosamine solution (184 mg/kg). Patients will be scanned twice during the same MRI session, before and 2 hours after taking glucosamine orally. In addition to the CEST scans with GlcN, patients will undergo MRI scans with the standard contrast agent of gadolinium. This procedure will be done following the CEST scan. The CEST scan takes a few minutes (up to 10 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Women with suspicious finding/process in the breast that requires MRI examination
2. Age: Over 18 years.
3. For 10 patients of control group - patients without breast tumor, carriers of mutations in P53, BRCA2, BRCA1 or PTEN genes or women after genetic counseling who have been defined as having a 20% risk of developing breast cancer and are undergoing routine MRI.

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Sensitivity to glucosamine and / or gadolinium.
3. Renal failure with creatinine clearance less than 30 cc per minute.
4. Weight over 130 kg.
5. Patients who have undergone breast surgery in the past year.
6. Claustrophobia.
7. Cardiovascular instability, symptomatic heart disease, pacemaker, artificial heart valve.
8. Intra-body injection device.
9. A generalized (idiopathic) epileptic seizure that is pharmacologically unbalanced.
10. Metabolic instability (water economy, electrolytes, sugar).
11. Suffers from a gastrointestinal disorder that affects absorption.
12. Fever or evidence of a microbiological contaminant.
13. Women using drugs that are related to derivatives of warfarin-coumadin.
14. Women with phenylketonuria
15. Inability to sign informed consent.
16. COVID-19

In addition, all examinees will be subject to the accepted criteria for inclusion and exclusion of the MRI unit at Meir Medical Center.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection and diagnosis of malignant tumors in the breast | up to three years (MRI scans and data collection and interpretation will last up to 2 years; post processing, reports and publications will last about one more year)
  Detection and diagnosis of malignant tumors in the breast without the use of gadolinium contrast agent.
  The proposed GlcN CEST MRI method is based on the ability of tumors to accumulate glucosamine in a preferred manner (Warburg effect). Therefore, the new method allows the acquisition of new information that is not obtained by other imaging methods: the method allows the presentation of a new contrast image in MRI that expresses metabolic changes in the tumor, expressed as % GlcN CEST.

SECONDARY OUTCOMES:
Tumor classification: benign or malignant | 3 years (data collection and post processing)
  It is hypothesized that the proposed study will allow to distinguish between malignant and benign tumors based on the quantification of glucosamine and its metabolites uptake in the tumor. Tools for assessing this outcome measure:
  Construction of a CEST scale bar based on magnetization transfer asymmetry ratio (MTRasym) maps that will be evaluated on a predetermined scale (expressing the effect as %).
  A GlcN signal rising over or equivalent to the MTRasym impact of 3% will be considered as a success metric for malignant tumors. MTRasym percentages are expected to be minimal to zero in benign tumors because GlcN uptake is likely to be poor.
Glucosamine CEST scale bar | Three years (data collection and post processing)
  Create a scale bar representing the CEST intensity (percent) in the tumor, which will be used to determine the degree of malignancy.
Finding correlation between research results and selected pathological parameters to better identify breast cancer | 3 years (data collection and statistical evaluation)
  In order to examine and/or assess the correlation between disease manifestation and the GlcN CEST MRI finding, the research results will be compared to selected pathological/ histopathological parameters of the patients (such as disease classification, grade, presence of estrogen receptors, progesterone receptor status, HER2, Ki-67 status, and so on). The statistical significance of the correlation will be assessed
Using Mathematical model | up to 3 years (post processing-1 year)
  As glucosamine accumulates in tumors, the level of malignancy and activity of distinct regions in the tumor can be assessed using mathematical modeling of the numerous products that contribute to the CEST MRI signal.
  To resolve individual contributions to the GlcN CEST effect, the Z spectra will be analyzed using a multi-pool Gaussian fitting model for the separation of the water, Magnetization transfer (MT), hydroxyl, amine/amide, and Nuclear Overhauser enhancement (NOE) signals.
  The fitting of the Z-spectrum to the sum of multiple Gaussian functions will be performed using the following equation: y= iAiexp [ -4ln2(x-ωi)2 / σi2] where ω is the frequency offset from the water resonance (ppm), and Ai, ωi and σi are the amplitude, frequency offset (ppm) and linewidth (ppm) of the CEST peak for the ith proton pool, respectively. Thus, using the multi-pool Gaussian fitting approach will enable to account for the contribution of each metabolite to the total GlcN CEST effect.